CLINICAL TRIAL: NCT02572414
Title: Health Promotion for HIV Positives: A Randomized Trial With HIV Positive Black Men
Brief Title: Men Together Making a Difference: Health Promotion for Black Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 813202; R01MD006232 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2015-10-08 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: HIV; Cardiovascular Disease; Diabetes; Hypertension; Colon Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hypertension; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Promotion Intervention (Experimental): Men Together Making a Difference Health Promotion Intervention consisted of three, 3-hour weekly small-group intervention sessions led by a trained facilitator using a detailed, scripted manual designed to increase adherence to guidelines for physical activity, 5-a-Day diet, and colon cancer screening.
  Interventions: Behavioral: Health Promotion Intervention
- Health Awareness Control (Active Comparator): Health Awareness Control Intervention consisted of one 1-hour small-group session led by a trained facilitator. Participants viewed and discussed video clips on physical activity, fruit and vegetable consumption, and colon cancer screening.
  Interventions: Behavioral: Health Awareness Control Intervention

INTERVENTIONS:
Behavioral: Health Promotion Intervention — Men Together Making a Difference Health Promotion Intervention, which included three, 3-hour weekly sessions, implemented in small groups by trained facilitators using scripted manuals, was designed to increase self-efficacy, outcome expectancy, and skills for behaviors tied to cardiovascular disease, diabetes, hypertension, and cancer. It encouraged men to adhere to guidelines for physical activity, 5-a-Day diet, and colon cancer screening. It encouraged at least 30 min of moderate-intensity aerobic activity on 5 days or at least 20 min of vigorous-intensity aerobic activity on 4 days and muscle-strengthening activity on at least 2 days each week. Participants identified their personal barriers to engaging in the recommended behaviors and strategies for surmounting those barriers.
  Other Names: Men Together Making a Difference Intervention
  Arms: Health Promotion Intervention
Behavioral: Health Awareness Control Intervention — Health Awareness Control Intervention consisted of one 1-hour small-group session led by a trained facilitator. Participants viewed and discussed video clips on physical activity, fruit and vegetable consumption, and colon cancer screening.
  Other Names: Control Intervention
  Arms: Health Awareness Control

SUMMARY:
African American men infected with HIV are living longer and are acquiring the same chronic non-communicable diseases affecting the general population of African American men age 40 years and older. African American men have disproportionately high rates of cardiovascular disease, hypertension, diabetes, kidney disease, and cancer, particularly prostate and colon cancer, but HIV is associated with an increased risk for co-morbidity from these conditions, a risk heightened by not only HIV infection itself, but also its treatment with antiretroviral therapy (ART). The risk for many of these chronic diseases is tied to behavior: risk is increased by physical inactivity and unhealthful diet. Although the high risk for behavior-linked chronic diseases among HIV-positive individuals has been recognized, there is a lack of evidence-based interventions specifically tailored to their needs.

Hence, the broad objective of this research is to identify strategies to empower HIV positive African American men to engage in behaviors that reduce their risk of chronic diseases. This research will test the efficacy of a theory-based, contextually appropriate health promotion intervention in inducing positive changes in behaviors linked to risk of chronic diseases among HIV positive African American men age 40 years or older and will identify the theoretical variables that mediate its efficacy.

In a randomized controlled trial, African American HIV positive men age 40 or older who are receiving ART for HIV will be randomized to the Men Together Making a Difference Health Promotion Intervention, which consists of three, 3-hour weekly intervention sessions, or the 1 session Health Awareness Control Group. The Men Together Making a Difference Health Promotion Intervention is based on social cognitive theory and the reasoned action approach integrated with formative research. Data will be collected at baseline, immediately post, and 3, 6 and 12 months post intervention. The trial will test whether the Men Making a Difference Health Promotion Intervention increases self-reported physical activity compared with the Health Awareness Control Group.

DETAILED DESCRIPTION:
African Americans are heavily burdened with preventable and treatable diseases, including cardiovascular disease, stroke, hypertension, diabetes, HIV/AIDS, sexually transmitted diseases (STDs), and cancers. African Americans have the highest age-adjusted death rates for heart disease, cancer, diabetes, and HIV/AIDS compared with other Americans. The broad objective of this research is to identify strategies to empower African American men to engage in healthful behaviors in an effort to help eliminate health disparities. Specifically, this research addresses the urgent need for health promotion interventions targeting African American men who are living with HIV. Despite the high risk for cardiovascular disease and other behavior-linked diseases, including diabetes and certain cancers, no studies have developed and tested interventions to encourage behaviors to reduce risk of chronic disease in African American HIV positive men, a sub-group comprising the largest segment of people living with HIV in the US. Moreover, irrespective of race and sex, few studies have tested interventions to increase behaviors to reduce risk of chronic diseases in people living with HIV.

From 2005 through 2007, the estimated number of persons living with HIV rose steadily in the 37 states with confidential name-based HIV infection reporting. At the end of 2007, an estimated 580,371 persons in these states were living with HIV infection, including 48% who were African-American and 73% who were men. In 2008, African Americans accounted for 52% of all new diagnoses of HIV infection in the 37 states with confidential name-based reporting. The estimated rate of diagnoses of HIV was higher in African American men (132 per 100,000) than in White men (17 per 100,000), Hispanic men (52 per 100,000), and African American women (56 per 100,000). In Philadelphia, where this study will be conducted, two-thirds of the people living with HIV/AIDS were African American in 2008, two-thirds were male, and one-half were age 45 years or older.

Since antiretroviral therapy (ART) has been available, there has been durable suppression of HIV replication, prevention of AIDS-defining opportunistic infections and malignancies, and higher survival and life expectancy rates in people living with HIV. In the US, 67% of people living with HIV in 2007 were age 40 or older. Because of the aging of the HIV positive population, several chronic non-HIV-related conditions are becoming increasingly important in the clinical treatment of HIV. Several reviews have drawn attention to the prevention and control of chronic diseases, including diabetes mellitus and cardiovascular, liver, and kidney diseases, affecting people living with HIV. Mounting evidence suggests that both HIV disease and its treatment with ART can accelerate the risks for chronic diseases associated with aging, particularly cardiovascular diseases and diabetes mellitus. Studies indicate that as HIV-infected patients live longer, they increasing experience mortality from causes not directly attributable to HIV. For instance, among people with HIV, the proportion of deaths not directly attributable to HIV increases with age from 36% among 30-year olds to 53% among 40-year olds and 72% among 50-year olds.

Quite apart from HIV infection, African Americans have higher mortality rates for cardiovascular disease, cerebrovascular diseases, and diabetes than do Whites. Some evidence also suggests that rates of hypertension and kidney disease are higher among HIV-infected African Americans than among HIV-infected Whites. Indeed, in a cohort study, the incidence of end-stage renal disease in people without HIV or diabetes was 2.3 times higher among African Americans than Whites, in those with diabetes but no HIV it was 2.3 times higher among African Americans than Whites, whereas in those with HIV but no diabetes, it was 8.1 times higher among African Americans compared with Whites. African Americans also have the highest mortality rates and the shortest survival rates for most cancers of any racial/ethnic group in the US. The death rate from colon cancer, the third most common cancer among African Americans, has decreased over the past 15 years, but incidence and mortality rates are still disproportionately high among African Americans, particularly men. The colon cancer incidence in African American men was 1.21 times higher than in White men and 1.31 times higher than in African American women, and the mortality rate in African American men was 1.44 times higher than in White men and 1.42 times higher than in African American women. The poor survival rates for colon cancers in African American men are linked to later stage at diagnosis and less access to appropriate and timely treatment.

Studies have shown that regular physical activity or physical fitness is associated with reduced risk of early mortality, cardiovascular disease, diabetes mellitus, and colon cancer. Consuming fruits and vegetables is associated with a lower risk of cardiovascular disease and certain cancers, but only 35% of African Americans report consuming fruit the recommended 2 or more times per day and only 24% report consuming vegetables the recommended 3 or more times per day. These findings underscore the need for interventions to encourage physical activity and fruit and vegetable consumption among African Americans. Screening is important to detect diseases in the early stages, but African Americans are less likely than Whites to report being screened for colon cancer. Reinhold et al. found that, despite significantly more visits with their primary care provider, HIV-infected patients age 50 years or older were less likely to have ever been screened for colon cancer than age- and gender-matched HIV-negative controls, and Bini et al. reported that HIV-infected individuals have a higher prevalence of colonic neoplasms and develop advanced neoplasms at a younger age than do uninfected individuals.

Few studies have examined health behaviors among HIV positive individuals, and fewer still have tested the efficacy of interventions that target behaviors linked to chronic diseases. This research will address this gap in the literature. It will test whether a health promotion intervention increases physical activity and other healthful behaviors compared with a health-awareness control group. The participants will be HIV positive African American men age 40 years and older who are ART patients. Participants will be recruited through the Clinical Registry of the Penn Center for AIDS Research, AIDS clinics and service organizations, HIV care providers, advertisements in a local newspaper, and word of mouth from participants.

The study will utilize a randomized controlled trial design. Computer-generated random number sequences will be used to randomly assign the men to the Men Together Making a Difference Health Promotion Intervention or the Health Awareness Control Intervention. The theoretical basis of the Men Together Making a Difference Health Promotion Intervention is social cognitive theory and the reasoned action approach. The intervention will seek to increase self-efficacy, outcome expectancy, behavioral skills, and risk-reduction knowledge for behaviors linked to cardiovascular disease, hypertension, diabetes, and cancer, including physical activity, fruit and vegetable consumption, fat consumption, and colon-cancer screening. The intervention will help men assess their health behavior, identify personal barriers to engaging in the behaviors, develop strategies for surmounting those barriers, and gain support for behavior change.

Participants will complete assessments before the intervention, immediately post and 3, 6, and 12 months post-intervention. Self-report measures will be collected using audio computer-assisted self-interviewing. The primary outcome is a binary variable indicating whether the participant met the 2008 Department of Health and Human Services physical activity guideline of engaging in muscle-strengthening activity on 2 days and engaging in either 20 min of vigorous-intensity activity on at least 4 days or 30 min of moderate-intensity activity on at least 5 days in the previous 7 days. The study tests whether the Men Together Making a Difference Health Promotion Intervention increases adherence to physical activities guidelines during the post-intervention period compared with the Health Awareness Intervention control group and whether social cognitive theory and reasoned action approach variables mediate the effects of the intervention.

A power analysis was used to calculate the sample size needed to detect a clinically significant difference in adherence to physical activity guidelines of 9.1 percent, a relative increase of 58.0%. Based on the sample of HIV positive men age 40 or older in Project Eban, estimated correlation among physical activity guideline adherence rates at 3-, 6-month, and 12-month follow-up is intraclass correlation (ICC) = 0.314. Assuming a 2-tailed test, alpha = 0.05, ICC = 0.314, 20% attrition, and a 9.1% increase in physical activity guideline adherence from 15.7% in the control group to 24.8% in the health promotion intervention group, a total N of 384 men enrolled will yield statistical power of 0.82.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older
* Self-identify as Black or African American
* Receiving ART for HIV

Exclusion Criteria:

* Blood pressure of 180/110 mm Hg or higher
* Plan to relocate beyond a reasonable distance from the study in the next 18 months or do not have an address where they can receive mail
* Participated in any health promotion intervention trial targeting physical activity, diet, or prostate or colon cancer screening in the past 12 months.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Adherence to Department of Health and Human Services physical activity guideline | up to 12 months post-intervention
  A binary variable indicating whether the participant met the 2008 Department of Health and Human Services physical activity guideline of engaging in muscle-strengthening activity on 2 days and engaging in either 20 min of vigorous-intensity activity on at least 4 days or 30 min of moderate-intensity activity on at least 5 days in the previous 7 days.

SECONDARY OUTCOMES:
Weighted average physical activity | up to 12 months post-intervention
  The weighted average physical activity is calculated by averaging days of vigorous and moderate aerobic activity, giving the average a weight of 5 and the days of strength building activity a weight of 2, taking the sum, and dividing the sum by 7.
Adherence to 5-a-Day diet guideline | up to 12 months post-intervention
  A binary variable indicating whether the participant met the 5-a-Day guideline of consuming at least 5 servings of fruit and vegetables daily in the previous 30 days

CONTACTS AND LOCATIONS:
Overall Officials: John B Jemmott III, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States